CLINICAL TRIAL: NCT01341912
Title: Clinical Study to Investigate the Long-Term Efficacy, Safety and Immunogenicity of Human-cl rhFVIII in Previously Treated Patients With Severe Haemophilia A - Extension Study to GENA-01
Brief Title: Study to Investigate the Long-term Efficacy and Safety of Human-cl rhFVIII in Previously Treated Patients (PTPs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENA-11
Record Dates: First submitted 2011-04-22; First posted 2011-04-26 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human-cl rhFVIII (Experimental): Recombinant FVIII derived from a human cell line.
  Interventions: Biological: Human-cl rhFVIII

INTERVENTIONS:
Biological: Human-cl rhFVIII — Human-cl rhFVIII is administered intravenously on demand for bleeding episodes and prophylactically in case of surgery. The dosage depends on the severity of the bleeding episodes and the surgery.

SUMMARY:
The purpose of the study is to study the long-term efficacy, safety and tolerability of Human-cl rhFVIII in previously treated patients with severe hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Completion of GENA-01 study with at least 50 Exposure Days (EDs) and at least 6 months study participation and immediate enrollment into GENA-11

Exclusion Criteria:

* Development of FVIII inhibitors (<=0.6 BU), during the course of the GENA-01 study
* Development of any severe liver or kidney disease (ALT and AST level > 5 times of upper limit of normal, creatine >120 micro mol/L) during the course of the GENA-01 study

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Georgetown University, Washington D.C., District of Columbia, United States
- Haematological Hospital SHAT "Joan Pavel", Sofia, Bulgaria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to all patients who had completed the GENA-01 study with at least 50 exposure days after at least 6 months of study participation (EU patients) or at least 15 months of study participation (US patients). Overall 21 patients were eligible for this study but only 3 patients decided to participate in this extension study.
Groups:
- Human-cl rhFVIII: Recombinant FVIII derived from a human cell line.
  Human-cl rhFVIII : Human-cl rhFVIII is administered intravenously on demand for bleeding episodes and prophylactically in case of surgery. The dosage depends on the severity of the bleeding episodes and the surgery.
Period: Overall Study
Arm/Group | Human-cl rhFVIII
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  Bulgaria | 3

OUTCOME MEASURES:

1. Primary Outcome: Long-term Immunogenicity
Description: Patients will be monitored for inhibitors against FVIII every 3 months. Blood samples were drawn and inhibitor activity was determined by the modified Bethesda assay (Nijmegen modification) in the central lab.
Time Frame: up to 3 years
Measure: Number; unit: occurrence of inhibitors
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 3
occurrence of inhibitors | 0

2. Secondary Outcome: To Determine Long-term Efficacy of Human-cl rhFVIII in the Treatment of Bleeding Episodes and in Surgical Prophylaxis
Description: The efficacy of human-cl rhFVIII will be determined using a 4 point efficacy assessment scale.
  After each infusion of IMP and at the end of a BE, the following efficacy assessment is made by the subject (together with the Investigator in case of on-site treatment):
  Excellent: Abrupt pain relief and/or unequivocal improvement in objective signs of bleeding within approximately 8 hours after a single infusion.
  Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 - 12 hours after an infusion requiring up to 2 infusions for complete resolution.
  Moderate: Probable or slight beneficial effect within approximately 12 hours after the first infusion requiring more than two infusions for complete resolution.
  None: No improvement within 12 hours, or worsening of symptoms, requiring more than 2 infusions for complete resolution.
  The assessment was made at the end of a BE in case more than one infusion was needed.
Time Frame: up to 3 years
Measure: Number; unit: percentage of bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 3
Number analyzed (Bleeding episodes) | 64
percentage of bleeding episodes
  Excellent | 71.88
  Good | 26.56
  Moderate | 1.56
  None | 0

ADVERSE EVENTS:
Time Frame: Patient 1 = 91 days Patient 2 = 57 days Patient 3 = 93 days
Arm/Group | Human-cl rhFVIII
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Only 3 patients participated in the study and all 3 patients withdrew consent prematurely. Therefore the results are summarized descriptively only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period